CLINICAL TRIAL: NCT00765778
Title: Mastering Hospital Antimicrobial Resistance and Its Spread Into the Community:the Role of Family Members and Caregivers in Dissemination of MDR in Rehabilitation Centers
Brief Title: Mastering Hospital Antimicrobial Resistance and Its Spread Into the Community
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: yehuda carmeli, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-YC-249-CTIL
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Bacterial Infection
Keywords: resistant bacteria rehabilitation centers
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Detailed activity:

* Family members and caregivers of carrier residents will be screened for ESBL and MRSA. Screening will be performed by obtaining nares and perirectal cultures. Nares cultures will be obtained by ward staff or research personnel who are experienced in performing this activity: a moisture swab will be applied gently to the distal part of both nares. Perirectal cultures, will be taken by swab, who will be applied to the perirectal area, either by staff as mentioned above, or will be given to the participants to perform by himself (with explanation on how to perform it).
* The Family and Caregiver Screening Form will be filled out; results of screening will be added to the forms. This data will be stored after removal of all Family members' identifiers for further analysis.
* In order to allow follow up, a list linking between the Family members' study number and his identifying details will be kept separately in the rehabilitation center. This list will not be transferred elsewhere.

DETAILED DESCRIPTION:
Detailed activity:

* Family members and caregivers of carrier residents will be screened for ESBL and MRSA. Screening will be performed by obtaining nares and perirectal cultures. Nares cultures will be obtained by ward staff or research personnel who are experienced in performing this activity: a moisture swab will be applied gently to the distal part of both nares. Perirectal cultures, will be taken by swab, who will be applied to the perirectal area, either by staff as mentioned above, or will be given to the participants to perform by himself (with explanation on how to perform it).
* The Family and Caregiver Screening Form will be filled out; results of screening will be added to the forms. This data will be stored after removal of all Family members' identifiers for further analysis.
* In order to allow follow up, a list linking between the Family members' study number and his identifying details will be kept separately in the rehabilitation center. This list will not be transferred elsewhere.
* Providing results to family members: results of screening will be / will not be reported to the participant (family member) based on local decision in each center.

ELIGIBILITY:
Inclusion Criteria:

* Family members or caregivers of patient hospitalized in rehabilitation center and who is known carrier of the target resistant population.
* Participating member older than 18 years, who attend the patient at least once a week, will be eligible for inclusion.

Exclusion Criteria:

* Age 18 years or less, attending the patient less than once a week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family members or caregivers of patient hospitalized in rehabilitation centers and who is known carrier of the target resistant population.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Family members and caregivers carriers of patients who are carriers of resistant bacteria /Family members and caregivers of patients who are carriers of resistant bacteria | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda carmeli, MD, Principal Investigator — TASMC
Locations (1):
- Tasmc, Tel Aviv, Israel

REFERENCES:
- [Background] Gottesman T, Agmon O, Shwartz O, Dan M. Household transmission of carbapenemase-producing Klebsiella pneumoniae. Emerg Infect Dis. 2008 May;14(5):859-60. doi: 10.3201/eid1405.071340. No abstract available. PMID 18439387